CLINICAL TRIAL: NCT02744222
Title: An International Multicenter Double-blind Placebo-controlled Randomized Study to Compare the Efficacy, Safety and Tolerability of BCD-054 (JSC BIOCAD, Russia), 180 μg and 240 μg, Versus Avonex® (Biogen Idec Ltd., UK) in Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Comparative Clinical Trial to Evaluate Efficacy, Safety and Tolerance of BCD-054 and Avonex® for Treatment of Patients With Remitting-relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCD-054-2
Record Dates: First submitted 2016-04-03; First posted 2016-04-20 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — sampeginterferon beta-1a; Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BCD-054, 180 mcg, biweekly (Experimental): Patients of Groups 1 will receive blinded BCD-054 180 mcg intramuscularly once every two weeks for the first 52 weeks (including a 4-week titration phase from Week 0 to Week 3 inclusive). Between every two injections of the active drug, once every 2 weeks, patients will receive intramuscular injections of placebo.From Week 53 until Week 100, patients of Groups 1 will receive open-label BCD-054 180 mcg or 240 mcg intramuscularly once every 2 weeks
  Interventions: Biological: BCD-054 180 mcg
- BCD-054, 240 mcg, biweekly (Experimental): Patients of Groups 2 will receive blinded BCD-054 240 mcg intramuscularly once every two weeks for the first 52 weeks (including a 4-week titration phase from Week 0 to Week 3 inclusive). Between every two injections of the active drug, once every 2 weeks, patients will receive intramuscular injections of placebo.From Week 53 until Week 100, patients of Groups 2 will receive open-label BCD-054 180 mcg or 240 mcg intramuscularly once every 2 weeks
  Interventions: Biological: BCD-054 240 mcg
- Avonex®, 30 mcg, weekly (Active Comparator): Patients of Group 3 (reference group) will receive blinded Avonex® 30 mcgintramuscularly once a week for the first 52 weeks (including a 4-week titration phase from Week 0 to Week 3 inclusive).
  Interventions: Biological: Avonex®
- Placebo, 0,5 ml, weekly (Placebo Comparator): Patients of Group 4 (placebo) will receive blinded placebo once a week for the first 20 weeks (including a 4-week titration phase from Week 0 to Week 3 inclusive)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BCD-054 180 mcg — 180 mcg intramuscularly once every two weeks
  Other Names: pegylated interferon beta-1a
  Arms: BCD-054, 180 mcg, biweekly
Biological: Avonex® — 30 mcg intramuscularly once a week
  Other Names: interferon beta-1a
  Arms: Avonex®, 30 mcg, weekly
Biological: BCD-054 240 mcg — 240 mcg intramuscularly once every two weeks
  Other Names: pegylated interferon beta-1a
  Arms: BCD-054, 240 mcg, biweekly
Other: Placebo — intramuscularly once a week (0,5 ml)
  Arms: Placebo, 0,5 ml, weekly

SUMMARY:
An International Multicenter Double-blind Placebo-controlled Randomized Study to Compare the Efficacy, Safety and Tolerability of BCD-054 (JSC BIOCAD, Russia), 180 μg and 240 μg, versus Avonex® (Biogen Idec Ltd., UK) in Patients with Relapsing-remitting Multiple Sclerosis

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study;
2. Men and women aged from 18 to 60 years (inclusive) on the day of signing informed consent;
3. Confirmed diagnosis of relapsing-remitting multiple sclerosis (according to McDonald criteria 2010) ;
4. Documentary evidence that within the last 12 months before signing informed consent the patient had:

   1. At least 1 relapse, or
   2. At least 1 Gadolinium enhancing T1-weighted lesion or 1 new T2-weighted lesion in dynamics.
5. The patient should be neurologically stable during 30 days before signing informed consent (i.e. the patient should not have any new or aggravated neurological symptoms, as told by the patient); or the patient's condition should be completely stabilized since the last relapse, and the duration of stabilization should be at least 30 days) ;
6. Patients of childbearing potential and their partners with preserved reproductive function must implement reliable contraceptive methods starting from signing informed consent to 4 weeks after the last dose of study therapy. This requirement does not apply to patients after operative sterilization. Reliable contraception methods include one barrier method in combination with one of the following: spermicides, intrauterine device/oral contraceptives;
7. Total EDSS score of 0 to 5.5 inclusive (assessed by the Assessing Neurologist).

Exclusion Criteria:

1. Primary or secondary progressive MS;
2. Other conditions (except for multiple sclerosis) that can affect the assessment of MS symptoms: to mask, aggravate, change symptoms of multiple sclerosis, result in clinical signs or laboratory instrumental findings suggesting multiple sclerosis;
3. A relapse during the screening period ;
4. Any acute infections, relapses of chronic infections or any other chronic diseases that are present on the day of signing informed consent and can, as judged by the Investigator, negatively affect the patient's safety during the study treatment;
5. HIV, hepatitis B, hepatitis C, or syphilis ;
6. Metabolic abnormalities (disorders) manifesting as:

   1. baseline creatinine levels increased more than 2-fold vs. upper limit of normal;
   2. baseline urea levels increased more than 3-fold vs. upper limit of normal;
   3. baseline ALT, AST or GGT levels increased more than 2.5-fold vs. upper limit of normal;
   4. baseline bilirubin levels increased more than 1.5-fold vs. upper limit of normal;
7. Baseline leukocyte counts lower than <3.0 × 109/L, platelet counts lower than <125 × 109/L or hemoglobin levels <100 g/L;
8. A history of severe depression, suicidal thoughts or suicide attempts ;
9. Signs of clinically significant depression (baseline Beck's score of more than 15);
10. A history of hypothyroidism/hyperthyroidism and/or baseline abnormalities of TSH levels vs. lower or upper limits of normal;
11. Epilepsy;
12. Pregnancy, lactation or planned pregnancy over the entire study period;
13. A history of use:

    * any time before signing informed consent: disease-modifying interferon beta drugs (interferon beta-1a, interferon beta-1b),
    * within 30 days before signing informed consent: glatiramer acetate;
    * within 6 months before signing informed consent: monoclonal antibodies, cytotoxic and/or immunosuppressive drugs, including but not limited to mitoxantrone, cyclophosphamide, cyclosporine, fingolimod, cladribine; or total lymphoid irradiation;
14. Systemic (i.v. or oral) corticosteroids used within 30 days before signing informed consent;
15. A history of intolerance of or allergy to pegylated proteins, interferon beta or other ingredients of BCD-054/Avonex®;
16. Known alcoholic or drug dependency or signs of present alcoholic/drug dependence that, in the Investigator's opinion, can be contraindications for study therapy of multiple sclerosis with interferon beta-1a or limit treatment compliance;
17. Inability to follow the Protocol procedures (in the Investigator's opinion).
18. Contraindications to MRI or use of gadolinium-containing contrast agents:

    1. Metal foreign objects in the body: magnetic implants, ferromagnetic clips for cerebral vessels, artificial heart valves, electronic middle ear implants, pacemakers;
    2. A history of allergy to gadolinium or gadolinium-containing contrast agents;

    с) Fear of cramped spaces; d) Kidney function impairment with a risk of delayed gadolinium elimination (creatinine level increased to more than 2 x upper limit of normal); e) Documented diagnosis of sickle cell or hemolytic anemia, hemoglobinopathy.
19. Any malignancies or a history of malignancies, except for cured basal cell carcinoma or cervical cancer in situ;
20. Vaccination within 4 weeks before signing informed consent (as told by the patient);
21. Participation in other clinical studies within 90 months before signing informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 399 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Time to first relapse after 52 weeks of blinded treatment with BCD-054 or Avonex | Week 52
  Time to first relapse after 52 weeks of blinded treatment with BCD-054 or Avonex

SECONDARY OUTCOMES:
CUA | Week 20, Week 52, Week 104
Proportion of patients without contrast-enhancing lesions | Week 20, Week 52, Week 104
Number of new or enlarging T2-weighted lesions | Week 20, Week 52, Week 104
Proportion of patients without new or enlarging T2-weighted lesions | Week 20, Week 52, Week 104
Changes in T2-weighted lesion volume | Week 20, Week 52, Week 104
Changes in hypointense T1-weighted lesion volume | Week 20, Week 52, Week 104
Annual average frequency of relapses | Week 20, Week 52, Week 104
Proportion of relapse-free patients | Week 20, Week 52, Week 104
Proportion of patients with sustained disability progression | Week 20, Week 52, Week 104
Expanded Disability Status Scale (EDSS) | Week 20, Week 52, Week 104
Timed 25-Foot Walk | Week 20, Week 52, Week 104
9-Hole Peg Test (9 HPT) | Week 20, Week 52, Week 104
Symbol Digit Modalities Test (SDMT) | Week 20, Week 52, Week 104
The proportion of patients who developed AEs/SAEs that, in the Investigator's opinion, are related to BCD-054 or Avonex® | Week12, Week 20, Week 52, Week 104
The proportion of patients, in each group, who developed СТСАЕ v. 4.03 Grade 3-4 AEs that, in the Investigator's opinion, are related to BCD-054 or Avonex® | Week12, Week 20, Week 52, Week 104
The proportion of patients, in each group, who discontinued the study due to AEs/SAEs | Week12, Week 20, Week 52, Week 104
The proportion of BAb- and NAb-positive patients | Week 20, Week 52, Week 104
AUC (0-168 hours) | from 0 to 168 hours after the first full dose of BCD-054 or Avonex® (Week 4)
  Area under the IFN-β1а concentration vs. time curve to 168 h (AUC(0-168)) with the first full dose of BCD-054 or Avonex® (Week 4)
AUC (0-336 hours) | from 0 to 336 hours after the first full dose of BCD-054 or Avonex® (Week 4)
  Area under the IFN-β1а concentration vs. time curve to 336 h (AUC(0-336)) with the first full dose of BCD-054 or Avonex® (Week 4)
AUCss (0-168 hours, 0-336 hours) | from 0 to 168 hours and from 0 to 336 hours since the introduction of 17 injections
  AUCss (0-168 hours, 0-336 hours) - area under curve "concentration - time" from 0 to 168 hours and from 0 to 336 hours(since the introduction of 17 injections, in steady state conditions)
AUECss (0-168 hours, 0-336 hours) | from 0 to 168 hours and from 0 to 336 hours after isince the introduction of 17 injections
  AUECss (0-168 hours, 0-336 hours) - area under effect curve "concentration of MxA-protein/neopterin - time" from 0 to 168 hours and from 0 to 336 hours (since the introduction of 17 injections, in steady state conditions)
AUEC (0-168 hours) | from 0 to 168 hours after the first full dose of BCD-054 or Avonex® (Week 4)
  Area under the effect (concentration of MxA protein/neopterin) vs. time curve to 168 h (AUC(0-168)) with the first full dose of BCD-054 or Avonex® (Week 4
AUEC (0-336 hours) | from 0 to 336 hours after the first full dose of BCD-054 or Avonex® (Week 4)
  Area under the effect (concentration of MxA protein/neopterin) vs. time curve to 336 h (AUEC(0-336)) with the first full dose of BCD-054 or Avonex® (Week 4)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JCS BIOCAD
Locations (1):
- State Budgetary Healthcare Institution of Nizhny Novgorod region " "Regional Clinical Hospital N.A. Semashko, Nizhny Novgorod", Nizhny Novgorod, Russia

IPD SHARING:
Plan to Share IPD: No